CLINICAL TRIAL: NCT06755047
Title: 3D Ultrasound Placental Volume and Vascular Indices Versus 2D Parameters for Diagnosis of Placenta Accreta Spectrum
Brief Title: 3D Placental Volume in Placenta Accreta
Status: Recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Mohamed Gamal M.fekry, Lecturer obstetric and gynecology, Specialist Urogynecology, Assiut University
Other Study IDs: 3D
Record Dates: First submitted 2024-12-12; First posted 2025-01-01 (Actual); Last update posted 2025-01-01 (Actual); Status verified 2024-12

CONDITIONS: Placenta Accreta
MeSH Terms: conditions — Placenta Accreta

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- 3D Ultrasound: 3D ultrasound placental volume, vascularization index, flow index and VF index
  Interventions: Radiation: 3D Ultrasound
- 2D ultrasound: lacunar vascular flow, abnormal utero-placental interference, myometrial thinning (>1mm), absence of the retroplacental myometrium, interruptions or irregularities at the level of the utero-vesical interference, lower uterine segment hypervascularity
  Interventions: Radiation: 2D ultrasound

INTERVENTIONS:
Radiation: 3D Ultrasound — 3D placental volume and vascular indices
  Groups: 3D Ultrasound
Radiation: 2D ultrasound — 2D placental criteria of invasion and color Doppler
  Groups: 2D ultrasound

SUMMARY:
Placenta Accreta spectrum is a major obstetric disease nowadays. Different methods are used for antenatal diagnosis. In our study, investigators are aiming to compare 2 common ways for diagnosis, i.e; 3D Ultrasound and 2D with color Doppler.

DETAILED DESCRIPTION:
The word placenta accreta spectrum disorders (PASD) implies an atypical implantation of the placenta into the uterine wall and has been used to express placenta accreta, increta and percreta. Placenta accreta is a placenta where the placental villi sick on directly to the myometrium. Placenta increta is a placenta where the placental villi attack into the myometrium and placenta percreta is a placenta where the villi invade through the myometrium and into serosa. No antenatal diagnostic method gives the clinician 100% assurance of either ruling in or ruling out the existence of placenta accreta. The definitive diagnosis of placental accreta spectrum is frequently ended postpartum on hysterectomy specimens when an area of accretion shows chorionic villi which make direct contact with the myometrium and absence of deciduae. Antenatal ultrasound is the method of choice used to establish the diagnosis and direct clinical management.The combined use of power Doppler with three dimensional (3D) ultrasound provides the possibility of quantifying moving blood within a volume of interest. Three indices are calculated, namely vascularization index (VI), flow index and vascularization flow index

ELIGIBILITY:
Inclusion Criteria:

* pregnant women with placenta previa

Exclusion Criteria:

* congenital anomalies of placenta Placental separation Uterine anomalies

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Gender Based: Yes
Study Population: All patients with placenta previa from 24 -39 weeks will be counselled to participate in the study. Patients will be enrolled in one of the 2 groups. Group 1, 3D Ultrasound with placental volume and vascular indices will be calculated. Group 2 , 2D ultrasound parameters and color Doppler study will be performed.
Sampling Method: Non-Probability Sample
Enrollment: 38 (Estimated)
Dates: Start 2024-12-31 (Actual); Primary Completion 2025-04 (Estimated); Study Completion 2025-05 (Estimated)

PRIMARY OUTCOMES:
Vascular index | 1 months
  3D Vascularization index

SECONDARY OUTCOMES:
2D ultrasound | 1 months
  myometrial thinning (>1mm),

CONTACTS AND LOCATIONS:
Locations (1):
- Women's Health Hospital, Asyut, Egypt